CLINICAL TRIAL: NCT02261363
Title: A Mixed Method EMA Assessment of Cognition and Behavior Among New ENDS Users: An Observational Cohort Study
Brief Title: The Moment Study: Mixed Method E-cigarette Study
Acronym: Moment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Truth Initiative (Other)
Responsible Party: Principal Investigator, Jennifer Pearson, Research Investigator, Truth Initiative
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00008526
Record Dates: First submitted 2014-10-03; First posted 2014-10-10 (Estimated); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ecig group 1 (Experimental): On study day 6, we provided participants with two NJOY King 5-packs of cigalike e-cigarettes and asked them to take at least three puffs a day to ensure that they had some exposure to the product in the first week. On day 13, we gave participants two additional NJOY King 5-packs and instructed them to use or not use the e-cigarettes as they wished.
  Interventions: Other: Ecig group 1

INTERVENTIONS:
Other: Ecig group 1 — E-cigarettes were 3% nicotine and of tobacco or menthol flavor, depending on participants' usual flavor preference.

SUMMARY:
The universe of tobacco products is expanding, with new noncombustible products gaining popularity even as the reduction in prevalence of cigarette smoking slows or stalls. E-cigarettes, or Electronic Nicotine Delivery Systems (ENDS), are the most prevalent of these emerging noncombustible products. With sales increasing rapidly and more efficient pulmonary delivery devices under development, ENDS are likely to play an increasing role in the future tobacco market. Little is known about the cognitions and behaviors leading to or sustaining ENDS use. Smokers may use ENDS to subvert smoking restrictions, to reduce perceived smoking harms, or for smoking cessation. Evidence about ENDS use is emerging from national surveillance and laboratory research, but the majority of information on ENDS is limited to retrospective surveys and convenience samples of White male ENDS users. The investigators research suggests Black smokers are less likely than White smokers to try and be current ENDS users, perhaps due to a greater degree of perceived harm associated with ENDS, a preference for menthol, or cultural norms. Thus, it is timely and critical to study how all smokers, including Blacks and menthol smokers, experience and initiate ENDS use employing valid, innovative research methods.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

1. be aged 18 years or older
2. reside in Washington, D.C. metro area (including VA and MD suburbs)
3. be proficient in English
4. be daily smoker with at least 5 years of established daily smoking

   * A person will be categorized as a daily smoker if he reports daily smoking of at least 8 cigarettes a day for the past 5 years, and records an exhaled air carbon monoxide (CO) level > 8 parts-per-million (ppm) at the baseline in-person meeting.
   * Daily smokers will be eligible for the main study if they do not intend to quit in the next 30 days.
   * If they do intend to quit in the next 30 days, eligible daily smokers will be enrolled in the second arm of the study.
5. not taking smoking cessation medications;
6. smoked LCC/cigars/hookah less than 5 times in last 30 days
7. have not used other tobacco products in last 30 days
8. have not used an ENDS product (electronic cigarette) in the last 30 days
9. be interested in trying an ENDS
10. have an iPhone or Android that allows installation of applications and use it daily
11. have a phone plan that allows unlimited text messages
12. be willing to travel to the data collection cite four times in three weeks
13. not be breastfeeding or planning to become pregnant
14. not have heart disease/uncontrolled blood pressure
15. not have psychosis/suicidal thoughts
16. not be currently enrolled in an alcohol treatment program
17. not be out of town for more than 5 nights in the next 6 weeks

Exclusion Criteria:

* Individuals who do not satisfy the criteria above will not be eligible for this study.
* There will be no involvement of vulnerable populations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- American Legacy Foundation, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Harvey EJ, Rubin LF, Smiley SL, Zhou Y, Elmasry H, Pearson JL. Mobile Phone Ownership Is Not a Serious Barrier to Participation in Studies: Descriptive Study. JMIR Mhealth Uhealth. 2018 Feb 19;6(2):e21. doi: 10.2196/mhealth.8123. PMID 29459355
- [Derived] Pearson JL, Smiley SL, Rubin LF, Anesetti-Rothermel A, Elmasry H, Davis M, DeAtley T, Harvey E, Kirchner T, Abrams DB. The Moment Study: protocol for a mixed method observational cohort study of the Alternative Nicotine Delivery Systems (ANDS) initiation process among adult cigarette smokers. BMJ Open. 2016 Apr 22;6(4):e011717. doi: 10.1136/bmjopen-2016-011717. PMID 27105716

RESULTS

PARTICIPANT FLOW:
Groups:
- Ecig Group 1: On study day 6, we provided participants with two NJOY King 5-packs of cigalike e-cigarettes (3% nicotine; tobacco or menthol flavor, depending on participants' usual flavor preference) and asked them to take at least three puffs a day to ensure that they had some exposure to the product in the first week. On day 13, we gave participants two additional NJOY King 5-packs and instructed them to use or not use the e-cigarettes as they wished.
Period: Overall Study
Arm/Group | Ecig Group 1
Started | 117
Completed | 96
Not Completed | 21
Not completed — Lost to Follow-up | 21

BASELINE CHARACTERISTICS:
Groups:
- Ecig Group: This is an interventional study with one group.
Arm/Group | Ecig Group
Number analyzed (Participants) | 96
Age, Categorical [Count of Participants; unit: Participants] — self-reported age
  Participants
    <=18 years | 0
    Between 18 and 65 years | 96
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 92
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 65
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Menthol preference [Number; unit: participants] — self-reported menthol preference
  participants
    Menthol | 72
    non-menthol | 24
Educational attainment [Number; unit: participants] — self-reported education
  participants
    high school graduate or lower | 30
    some college or more | 66
Fagerstrom test [Number; unit: participants] — Fagerstrom score is a self-reported measure of cigarette dependence. Lower scores equate to lower levels of nicotine dependence, with less than or equal to 5 equating to low dependence, 6-7 equating to moderate dependence, and 8-10 equating to high dependence.
  participants
    <=5 | 16
    6-7 | 57
    8-10 | 23
Age of first cigarette [Number; unit: participants] — self reported age when first tried cigarettes
  participants
    <=14 years | 31
    15-18 years | 48
    19-24 years | 12
    25-55 years | 5

OUTCOME MEASURES:

1. Primary Outcome: Cigarette Use
Description: Change in the average number of cigarettes per day comparing average cigarettes per day on study day 6 (last day of cigarette-only use) to average cigarettes per day on study day 7 (first day of e-cigarette and cigarette use).
Time Frame: Study Day 7, Week 2
Measure: Mean (95% Confidence Interval); unit: cigarettes
Arm/Group | Ecig Group 1
Number analyzed (Participants) | 96
cigarettes | -1.82 [-2.32 to -1.32]

ADVERSE EVENTS:
Arm/Group | Ecig Group 1
Serious Adverse Events (participants affected / at risk) | 0/96
Other Adverse Events (participants affected / at risk) | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No